CLINICAL TRIAL: NCT06126367
Title: Assessment of Lipoprotein(a) and Endogenous Fibrinolysis in Atherosclerotic Cardiovascular Disease/Aortic Valve Disease
Acronym: ALFA
Status: Recruiting | Type: Observational
Sponsor: East and North Hertfordshire NHS Trust (Other Government)
Responsible Party: Principal Investigator, Prof Diana Gorog, Professor, University of Hertfordshire
Other Study IDs: RD2023-43
Record Dates: First submitted 2023-11-06; First posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Atherosclerosis; Aortic Valve Disease
Keywords: Lipoprotein (a); Global thrombosis test; Endogenous fibrinolysis
MeSH Terms: conditions — Atherosclerosis; Aortic Valve Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients identified as eligible for treatment with either a PCSK9i or inclisiran
  Interventions: Diagnostic Test: Thrombotic assessment; Diagnostic Test: Measurement of Lp(a)
- Patients with moderate or severe aortic calcification identified by non-enhanced cardiac CT scan
  Interventions: Diagnostic Test: Thrombotic assessment; Diagnostic Test: Measurement of Lp(a)

INTERVENTIONS:
Diagnostic Test: Thrombotic assessment — The Global Thrombosis Test (Thromboquest Limited, UK) is an in vitro method imitating high shear stress conditions akin to that which exist in a severely stenosed artery. The test measures platelet reactivity (occlusion time) and endogenous fibrinolysis time (lysis time).
  Thromboelastography is a technique that assesses the whole process of clotting and its viscoelastic properties, from the initial activation and aggregation of platelets, to the role of thrombin and finally the stability of the formed clot, as a measure of fibrinolytic resistance.
  Plasma will be stored for subsequent analysis of other thrombotic, fibrinolytic, inflammatory and coagulation markers as deemed appropriate.
  For patients deemed eligible for treatment with either a PCSK9i or inclisiran, this will be assessed prior to commencing treatment and also 3-6 months after starting treatment.
  This will only be assessed once for patients with moderate or severe aortic valve calcification.
Diagnostic Test: Measurement of Lp(a) — Lp(a) will be measured by particle enhanced immunotubidimetricassay. Human lipoprotein (a) agglutinates with latex particles coated with anti-Lp(a) antibodies. The precipitate is determined turbidimetrically at 800 / 660 nm. The platform employed will be the Roche® Immunoassay Analyser (Roche Diagnostics GmbH, Sandhofer Strasse 116, D-68305 Mannheim). Traceability: This method has been standardized against the IFCC (International Federation of Clinical Chemistry) reference material SRM2B for nmol/L.
  For patients deemed eligible for treatment with either a PCSK9i or inclisiran, this will be assessed prior to commencing treatment and also 3-6 months after starting treatment.
  This will only be assessed once for patients with moderate or severe aortic valve calcification.

SUMMARY:
Prior studies have shown that impaired endogenous fibrinolysis is a novel, independent cardiovascular risk factor in patients with myocardial infarction and there is currently no known chronic treatment to enhance endogenous fibrinolysis.

To date, no therapies have been able to sufficiently reduce Lp(a) and therefore it was considered to be a non-modifiable cardiovascular risk factor. New data, however, has shown that PCSK9 inhibitors and inclisiran (medication that you have been deemed eligible for in order to help further reduce your cholesterol levels) to reduce Lp(a) levels by approximately 20-25%.

The aim of this study to is to assess:

1. if there is an association between raised Lp(a) level in blood and the effectiveness of endogenous fibrinolysis (lysis time).
2. whether lowering Lp(a) with PCSK9i or inclisiran can enhance endogenous fibrinolysis

DETAILED DESCRIPTION:
The risk of a clot forming in a blood vessel, which can cause a heart attack or stroke, is determined partly by how "sticky" the blood is and partly by the effectiveness of the natural defences in the blood in dissolving any clots that start forming (clot lysis, or "fibrinolysis").

In the last few years, using new blood testing techniques, we and other groups, have shown that individuals who have less effective natural clot lysis, have a much higher risk of heart attack, stroke and death, even despite current best medications.

Therefore, we would like to find medications that can make clot lysis more effective, in such individuals, to reduce their risk of stroke and heart attack. Unfortunately, most blood thinning tablets for long term use do not improve clot lysis. Earlier, our group has shown that the anticoagulant apixaban, mildly improved clot lysis

Elevated concentration of Lp(a) in the blood is a risk factor for the development of cardiovascular disease including coronary artery disease and narrowing of the aortic valve. Lp(a) may exert its adverse effects by impairing fibrinolysis. Plasmin is an important enzyme present in blood that degrades many blood plasma proteins, including fibrin clots. Lp(a) has a high degree of homology to plasminogen (a pro-enzyme that is cleaved to form plasmin) and may cause thrombosis by competitively inhibiting t-PA-mediated plasminogen activation and tPA-mediated clot lysis. Furthermore, Lp(a) stimulates the activity of PAI-1, which is the major inhibitor of the fibrinolytic system.

Until recently, Lp(a) has been considered a non-modifiable cardiovascular risk factor as few therapies are available to sufficiently reduce Lp(a) levels. New data, however, have shown that novel cholesterol lowering treatments, namely PCSK9 inhibitors and inclisiran (a long-acting silencing RNA) can reduce Lp(a) levels by approximately 20-25%.

Given Lp(a) is a causal risk factor for cardiovascular outcomes, it is important to know if a reduction in Lp(a) can favourably modify endogenous fibrinolysis.

If Lp(a) level is directly related to the effectiveness of endogenous fibrinolysis, then medications that reduce Lp(a) (currently PCSK9i and/or inclisiran, and others in development) could be used as targeted treatment for patients who despite optimal antithrombotic therapy, demonstrate impaired endogenous fibrinolysis.

ELIGIBILITY:
Inclusion Criteria:

1) Male and female patients aged 18 years or over

2) i) Patients identified as eligible for treatment with either a PCSK9i or inclisiran ii) Patients diagnosed with moderate or severe calcific aortic stenosis based on non-enhanced Cardiac CT scan

3) Willing and able to understand the Participant Information Sheet and provide informed consent

4) The patient must agree to comply with the drawing of blood samples for the assessments

5) The patient does not meet any of the exclusion criteria

Exclusion Criteria:

1. Inability to provide valid informed consent
2. Male and female patients aged < 18 years of age
3. The patient has, in the opinion of the investigator, significant neurological, hepatic, renal, endocrine, gastrointestinal, pulmonary, haemorrhagic, metabolic or other disease likely to confound the study requirements or analyses
4. The patient has a history of substance abuse or demonstrates signs or clinical features of active substance abuse or psychiatric disease
5. Alcohol consumption above recommended safe levels (i.e., more than 14 units per week) due to the potential effects of high alcohol levels on platelet reactivity
6. Any illness deemed significant by the investigator during the four (4) weeks preceding the screening period of the study
7. Any major bleeding diathesis or blood dyscrasia (platelets < 70 x 109/l, Hb < 8 g/dl, INR > 1.4, APTT > x 2 upper normal limit, leucocyte count < 3.5 x 109/l, neutrophil count < 1 x 109/l)
8. Currently enrolled in an investigational device or non-licensed drug trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1) Male and female patients aged 18 years or over.
  2) i) Patients identified as eligible for treatment with either a PCSK9i or inclisiran ii) Patients diagnosed with moderate or severe calcific aortic stenosis based on non enhanced Cardiac CT scan
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Thrombotic status | 3-6 months
  Change in thrombotic status as measured by Lysis Time (LT) using the GTT from baseline to 6-months post initiation of PCSK9i or inclisiran
Lipoprotein(a) levels | 3-6 months
  Change in lipoprotein(a) levels from baseline to 6-months post initiation of PCSK9i or inclisiran

CONTACTS AND LOCATIONS:
Overall Officials: Diana A Gorog, MD, PhD, Principal Investigator — East and North Hertfordshire NHS Trust
Locations (1):
- East and North Herts NHS Trust, Stevenage, United Kingdom